CLINICAL TRIAL: NCT04702594
Title: Impact of Music Therapy on Psycho-behavioral Disorders of the Elderly Suffering From Neuro-cognitive Disorders
Brief Title: Music Therapy and Psycho-behavioral Disorders in the Elderly Population
Acronym: DEMUse
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 69HCL20_0489
Record Dates: First submitted 2021-01-07; First posted 2021-01-11 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Behavioral Disorder; Music Therapy
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- UHR and SRH (Experimental): All patients over the age of 60 present in the UHR and hospitalized in SRH with behavioral disorders in the context of a neurocognitive disorder
  Interventions: Behavioral: Music therapy session via tools validated by MUSIC CARE

INTERVENTIONS:
Behavioral: Music therapy session via tools validated by MUSIC CARE — Use of the MUSICARE tool, a digital space allowing access to different validated methods of music therapy. Music listening times are offered to patients with cognitive impairment with psycho-behavioral symptoms. The sessions are individual or group performed by a psychomotor therapist in UHR and volunteer caregivers trained in SRH. The sessions last on average 20-30min.

SUMMARY:
Since the 1990s, neuroscience, with functional MRI, has made it possible to understand the beneficial neurophysiological effect of music on man and his brain. They have shown that music stimulates brain plasticity and contributes to the reorganization of the affected neural circuits. The concept of cerebral plasticity and cerebral symphony have thus been developed. In March 2008, the HAS (High Authority for Health) proposed in its recommendations good practices concerning the management of neurodegenerative diseases that "Music therapy, aromatherapy, multisensory stimulation ... could improve certain of behavior's aspects ". Music has shown that memory capacity can remain present in people with Alzheimer's disease even in the advanced stages. Music also improves the well-being of patients with Alzheimer's or mixed dementia living in institutions and reduces the suffering of caregivers. It improves communication with others, including those who have lost the usual codes of communication and improves the quality of sleep of elderly people living in institutions.

However, although musical interventions have recently gained popularity as a non-pharmacological treatment for dementia, the scientific evidence warrants further research.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 60 present in the reinforced hospital unit during the study period
* Patients over 60 years hospitalized in follow-up care and rehabilitation with behavioral disorders in the context of a neurocognitive disorder

Exclusion Criteria:

* Unpaired deafness
* Refusal to participate

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2021-01-18 (Actual); Primary Completion 2021-08-18 (Estimated); Study Completion 2021-08-18 (Estimated)

PRIMARY OUTCOMES:
Evolution of the NeuroPsychiatric Inventory (NPI) scale | Baseline, once a week during study participation and at the end of the patient's participation in the study (1 month after inclusion)
  The improvement in psycho-behavioral symptoms will be assessed by the NPI score provided by the MUSIC CARE application carried out by a caregiver.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Pierre Garraud, Lyon, France